CLINICAL TRIAL: NCT06079372
Title: A Phase 3, Randomized, Open-label, Parallel-arm, Active-controlled, Multicenter Study to Evaluate Safety and Efficacy of ALXN1850 Versus Asfotase Alfa Administered Subcutaneously in Pediatric Participants (2 to < 12 Years of Age) With Hypophosphatasia (HPP) Previously Treated With Asfotase Alfa
Brief Title: Phase 3 Study of ALXN1850 in Pediatric Participants With HPP Previously Treated With Asfotase Alfa
Acronym: CHESTNUT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8590C00004; ALXN1850-HPP-303 (Other: Alexion Pharmaceuticals, Inc.)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; HPP; Asfotase Alfa; ALXN1850
MeSH Terms: conditions — Hypophosphatasia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALXN1850 (Experimental): Starting at Day 1 of the Randomized Evaluation Period participants will receive ALXN1850 for a total of 24 weeks. Participants will receive bodyweight dependent doses of either 20mg, 35mg or 50mg of ALXN1850 once q2w via SC injection. During Part A of the OLE Period, participants will have frequent visits over the first 24 weeks; Part B of the OLE Period participants will have visits every 9 months for up to approximately 108 weeks.
  Interventions: Drug: ALXN1850; Drug: asfotase alfa
- asfotase alfa (Experimental): Starting at Day 1 of the Randomized Evaluation Period, participants will receive asfotase alfa for a total of 24 weeks. Participants will receive 6 mg/kg/week of asfotase alfa via SC injection as either 2 mg/kg 3 times per week or 1 mg/kg 6 times per week. Part A of the OLE Period participants will have frequent visits over the first 24 weeks; Part B will have visits every 9 months for up to approximately 108 weeks.
  Interventions: Drug: asfotase alfa

INTERVENTIONS:
Drug: ALXN1850 — ALXN1850 will be administered via subcutaneous (SC) injection.
  Arms: ALXN1850
Drug: asfotase alfa — Asfotase alfa will be administered via SC injection.

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of ALXN1850 versus asfotase alfa in pediatric participants with HPP previously treated with asfotase alfa.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HPP documented in the medical records
* Presence of open growth plates by X-ray during Screening Period
* Tanner stage 2 or less during the Screening Period
* Must have been treated with 6 mg/kg/ week of asfotase alfa via SC injection administered as either 2mg/kg 3 times per week or 1 mg/kg 6 times per week for ≥ 6 months before Day 1. Note: participants currently treated with 9 mg/kg (eg, 3 mg/kg 3 times per week) will not be allowed in the study.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, neurological disorders, or any other disorders that are capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data as determined by the Investigator.
* Diagnosis of primary or secondary hyperparathyroidism
* Hypoparathyroidism, unless secondary to HPP
* Any new fracture within 12 weeks before Day 1 (excluding pseudofractures)
* Planned surgical intervention which may impact the results of study assessments (in the opinion of the Investigator) during the Randomized Evaluation Period
* History of allergy or hypersensitivity to any ingredient contained in asfotase alfa or ALXN1850
* Body weight < 10 kg during the Screening Period

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Baseline Through Day 169

SECONDARY OUTCOMES:
Radiographic Global Impression of Change (RGI-C) Score at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in Rickets Severity Score (RSS) at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in 6-Minute Walk Test (6MWT) at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in Percent Predicted 6MWT at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in Bruininks Oseretsky Test of Motor Proficiency, Second Edition (BOT2) Score at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169
Change from Baseline in Peabody Developmental Motor Scales, Third Edition (PDMS-3) Score at the end of the Randomized Evaluation Period (Day 169) | Baseline, Day 169

CONTACTS AND LOCATIONS:
Locations (21):
- United States (6):
  - Research Site, Hartford, Connecticut
  - Research Site, Baltimore, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, Durham, North Carolina
  - Research Site, Nashville, Tennessee
- Research Site, Mar del Plata, Argentina
- Research Site, South Brisbane, Australia
- Research Site, Ottawa, Ontario, Canada
- Japan (4):
  - Research Site, Bunkyō City
  - Research Site, Minatoku
  - Research Site, Suita-shi
  - Research Site, Yonago-shi
- Turkey (Türkiye) (5):
  - Research Site, Altındağ
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Erzurum
  - Research Site, Istanbul
- United Kingdom (3):
  - Research Site, Birmingham
  - Research Site, Manchester
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR